CLINICAL TRIAL: NCT00237965
Title: The Use of Mole Mapping Diagrams to Increase Skin Self Examination Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 00001402
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2005-10-13 (Estimated); Status verified 2004-05

CONDITIONS: Melanoma
Keywords: Skin Self Examination; Mole Mapping Diagram; Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Behavioral: Mole Mapping Diagram

SUMMARY:
This study aims to improve Skin Self-Examination accuracy by a simple cost effective intervention requiring participants to complete a mole-mapping diagram.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects above age 18 of any ethnicity will be enrolled in this study.

Exclusion Criteria:

* Subjects will be excluded from the study if they have significant skin disease which would not allow manipulation of their photographs consistent with the rest of the subjects.
* Since the study instructions are in English, Non-English speakers will be excluded.
* Those with co-morbidity sufficiently severe to prevent them from being able to perform a SSE will be excluded.
* In addition, those with cognitive impairment who are unable to give informed consent, or to understand the study instructions given to them, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Martin A Weinstock, MD, Ph.D, Principal Investigator — Veterans Affairs Medical Center Providence, RI